CLINICAL TRIAL: NCT01252641
Title: A Phase 1/2, Open Label, Single Infusion Study of Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases (SB-728-T) in HIV Infected Subjects
Brief Title: Study of Autologous T-cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases in HIV-Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-728-1002
Record Dates: First submitted 2010-11-29; First posted 2010-12-03 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: HIV; HIV Infection
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB-728-T (Experimental): Subjects will receive one intravenous infusion of SB-728-T
  Interventions: Biological: SB-728-T

INTERVENTIONS:
Biological: SB-728-T — Each infusion will be 5-30 billion modified CD4+ T-cells

SUMMARY:
This research study is being carried out to study a new way to possibly treat human immunodeficiency virus (HIV). The agent is called SB-728-T which are CD4+ T-cells obtained from an individual that are genetically modified at the CCR5 gene by Zinc Finger Nucleases. The CCR5 gene is required for certain types of HIV to enter into and infect T-cells. T cells are one of the white blood cells used by the body to fight HIV. The most important of these are called "CD4+ T-cells"

Some people are born without the CCR5 gene on their T-Cells. These people remain healthy and are resistant to infection with HIV. Other people have a low number of CCR5 genes on their T-cells and their HIV disease is less severe and is slower to cause disease (AIDS).

The purpose of this research study is to find out whether SB-728-T is safe to give to humans and find out how this affects HIV.

DETAILED DESCRIPTION:
Laboratory studies have shown that when CD4+ T-cells are modified with Zinc Finger Nucleases SB-728, HIV is prevented from killing the CD4+ T-cells. On the basis of these laboratory results, there is the potential that this may work in humans infected with HIV and improve their immune system by allowing their CD4+ T-cells to survive longer.

The new treatment to be studied will involve removing white blood cells from the blood that contain CD4+ T-cells. The extracted CD4+ T-cells are then genetically modified by the Zinc finger Nucleases to be resistant to infection by removing the CCR5 gene from the surface of the CD4+ T-cell where HIV enters the cell. Additional genetically modified cells are manufactured and then re-infused back into the individual. Researchers hope that these genetically modified cells will be resistant to infection by HIV and will be able to reproduce additional resistant CD4+ T-cells in your body.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* CD4+ T-cell count >500 cell per millimeter cubed (cells/mm3)
* CD4+ T-cell nadir of >400 cells/mm3
* HIV viral load >1,000 copies per milliliter (mL)

Exclusion Criteria:

* Any viral hepatitis
* Acute HIV infection
* HIV viral load >1,000,000 copies/mL
* Active or recent (prior 6 months) AIDS defining complication
* Any HIV medications within the past 12 weeks
* Cancer or malignancy that has not been in remission for at least 5 years with the exception of successfully treated basal cell carcinoma of the skin
* Current diagnosis of NYHA grade 3 or 4 congestive heart failure or uncontrolled angina or arrhythmias
* History of bleeding problems
* Use of chronic steroids in past 30 days
* Pregnant or breast feeding
* Active drug or alcohol abuse
* Serious illness in past 30 days
* Currently participating in another clinical trail or any prior gene therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of SB-728-T cells infusion in HIV-1 positive subjects | 12 months
  Evaluate the safety and tolerability of a single infusion of 5-30 billion SB-728-T cells in HIV-1 positive subjects

SECONDARY OUTCOMES:
Evaluate persistence of HIV as measured by HIV-1 RNA, | 12 months
Change in CD4+ T-cell count | 12 months
Persistence of SB-728-T in the peripheral blood | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Winson Tang, M.D., Study Director — Sangamo BioSciences, Inc.
Locations (4):
- United States (4):
  - UCLA CARE Center, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Quest Clinical Research, San Francisco, California
  - Orlando Immunology Center, Orlando, Florida